CLINICAL TRIAL: NCT05913583
Title: Correlation Between Exposure to Immune Checkpoint Inhibitors Before Liver Transplantation for Hepatocellular Carcinoma and Post-transplant Graft Rejection
Brief Title: Correlation Between Pre-transplant ICI Exposure and Post-transplant Graft Rejection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-224-01
Record Dates: First submitted 2023-05-24; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-04

CONDITIONS: Graft Rejection; Hepatocellular Carcinoma; Immunotherapy; Immune Checkpoint Inhibitor
Keywords: hepatocellular carcinoma; liver transplantation; Immune checkpoint inhibitor; Graft rejection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICI group: Recipients with exposure to immune checkpoint inhibitors before liver transplantation
  Interventions: Drug: Immune checkpoint inhibitor
- non-ICI group: Recipients without exposure to immune checkpoint inhibitors before liver transplantation

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Immune checkpoint inhibitors work by blocking checkpoint proteins from binding with their partner proteins. This prevents the "off" signal from being sent, allowing the T cells to kill cancer cells.One such drug acts against a checkpoint protein called CTLA-4. Other immune checkpoint inhibitors act against a checkpoint protein called PD-1 or its partner protein PD-L1.
  Other Names: Anti-PD-1; Anti-PD-L1; Anti-CTLA-4
  Groups: ICI group

SUMMARY:
Immune checkpoint inhibitors (ICIs) have revolutionized the treatment of advanced HCC. The combination of the ICI and other treatment regimens (Anti-VEGF, locoregional therapies et al) produced superior results in patients with advanced-stage HCC compared to those treated with traditional therapeutic regimens. Liver transplantation (LT) offers excellent long-term outcomes for certain patients with HCC. However, the immune-stimulating property of ICIs may lead to rejection and even graft loss, damping their use in treating HCC before liver transplantation. Therefore, it is worthwhile to explore the relationship between exposure to ICIs before LT and the incidence of graft rejection and rejection-related death or graft loss after LT.

DETAILED DESCRIPTION:
This will be a retrospective and observational study, which will analyze the correlation between the use of ICIs and incidences of graft rejection and rejection-related death or graft loss after LT in consecutive recipients with LT for HCC at the Organ Transplantation Center of Sun Yat-sen Memorial Hospital of Sun Yat-sen University.

The primary aim of this study is to analyze the correlation between pretransplant exposure to ICIs and incidences of graft rejection and rejection-related death or graft loss within 1 year after liver transplantation.

The secondary aim is to analyze the risk factors for graft rejection and to explore the correlation between ICI exposure and posttransplantation complication, such as incidences of early allograft dysfunction (EAD), bleeding, infection, biliary and vascular complications et al.

The exploratory aim is to identify potential biomarkers in predicting graft rejection, such as subsets of lymphocytes and cytokines et al.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent must be obtained prior to any data collection.
2. Patients must have pathologically or cytologically or by radiological criteria proven hepatocellular carcinoma based on the AASLD practice guidelines.
3. All patients receiving liver transplantation for HCC.

Exclusion Criteria

1. Cholangiocellular carcinoma, combined hepatocellular and cholangiocarcinoma, and other rare types of liver cancer that are confirmed by histology/cytology.
2. Patients with incomplete follow-up data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort study will be performed on consecutive HCC patients who underwent LT for HCC. The pretransplant parameters, such as AFP, tumor status, BMI, and etiology et al, as well as posttransplant parameters, such as graft rejection, EAD, hospital death et al, will be analyzed.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Graft rejection | 1 year
  In this study, rejection was be defined as the elevation of transaminase during the recovery of liver function after LT (transaminases should gradually return to normal levels) or suddenly abnormal elevations of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 times the upper limit that can be reversed by adjusting the immunosuppression regimen. Hepatic artery or portal vein thrombosis, drug toxicity or other factors should be excluded as the reason for liver function injury. Liver biopsies were not necessary for the diagnosis of rejection. The rejection activity index (RAI) was scored according to the Banff criteria to record the severity of acute rejection. An RAI score of 4-5 was defined as mild rejection, 6-7 was defined as moderate rejection, and 8-9 was defined as severe rejection.

SECONDARY OUTCOMES:
Graft loss | 1 year
  Rejection related graft loss
Hospital death | 1 year
  rejection related death
Early allograft dysfunction (EAD) | First 7 days after liver transplantation
  EAD is defined by the presence of one or more of the following: total bilirubin ≥ 10 mg/dL (171 μmol/L) or, INR ≥ 1.6 on day 7, and ALT/AST > 2,000 IU/L within the first 7 days

OTHER OUTCOMES:
CD4 to CD8 T cell ratio | 1 year
  The ratio of CD4 to CD8 T cells
pDC to mDC ratio | 1 year
  The ratio of plasmacytoid dendritic cells to myeloid dendritic cells

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Organ Transplantation Center, Sun Yat-sen Memorial Hospital, Sun Yat-sen University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwacha-Eipper B, Minciuna I, Banz V, Dufour JF. Immunotherapy as a Downstaging Therapy for Liver Transplantation. Hepatology. 2020 Oct;72(4):1488-1490. doi: 10.1002/hep.31234. No abstract available. PMID 32171041
- [Background] Tran NH, Munoz S, Thompson S, Hallemeier CL, Bruix J. Hepatocellular carcinoma downstaging for liver transplantation in the era of systemic combined therapy with anti-VEGF/TKI and immunotherapy. Hepatology. 2022 Oct;76(4):1203-1218. doi: 10.1002/hep.32613. Epub 2022 Jul 30. PMID 35765265
- [Background] Katariya NN, Lizaola-Mayo BC, Chascsa DM, Giorgakis E, Aqel BA, Moss AA, Uson Junior PLS, Borad MJ, Mathur AK. Immune Checkpoint Inhibitors as Therapy to Down-Stage Hepatocellular Carcinoma Prior to Liver Transplantation. Cancers (Basel). 2022 Apr 19;14(9):2056. doi: 10.3390/cancers14092056. PMID 35565184
- [Background] Llovet JM, Castet F, Heikenwalder M, Maini MK, Mazzaferro V, Pinato DJ, Pikarsky E, Zhu AX, Finn RS. Immunotherapies for hepatocellular carcinoma. Nat Rev Clin Oncol. 2022 Mar;19(3):151-172. doi: 10.1038/s41571-021-00573-2. Epub 2021 Nov 11. PMID 34764464
- [Derived] Pang L, Xu L, Chen Z, Liu Y, Ding T, Ye Y, Lu X, Gu G, Lin H, Wu W, Man K, Liu C. Short-term prognosis of recipients with pretransplant exposure to immune checkpoint inhibitors after liver transplantation for hepatocellular carcinoma: A retrospective cohort study. Liver Res. 2025 Mar 8;9(3):221-230. doi: 10.1016/j.livres.2025.03.001. eCollection 2025 Sep. PMID 41112510